CLINICAL TRIAL: NCT06218615
Title: Expanding Clinical Trial Awareness Among Black Communities Through Digital Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RG1124067; NCI-2024-00180 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020288 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Services Research (Experimental): Participants watch a culturally tailored decision aid video. Surveys are completed before and after the video.
  Interventions: Other: Educational Intervention (Video); Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention (Video) — Watch video
  Other Names: Fostering Opportunities in Research Using Marketing Strategies (FOR US)
Other: Survey Administration — Answer survey questions

SUMMARY:
Under-representation of patients from racial/ethnic minority groups in cancer clinical trials is a major barrier to health equity. Black patients are significantly less likely to be enrolled in clinical trials compared with non-Hispanic White (White) patients although they carry a disproportionate burden of cancer mortality, the shortest survival rates, and are more likely to be diagnosed at later stages. Further, medical mistrust and lack of awareness and complexity of clinical trials are barriers that reduce the likelihood of clinical trial participation. The objective of this pilot study is to understand the effect of a culturally tailored decision aid (previously developed by our research team) on 1) medical mistrust, 2) patient knowledge about clinical trials, and 3) decision-making self-efficacy and determine the acceptability of the decision aid among Black patients currently or ever been diagnosed with cancer.

DETAILED DESCRIPTION:
This study will be conducted online through Qualtrics.

Participants will answer pre-test survey questions, watch the culturally tailored decision aid video [Fostering Opportunities in Research Using Marketing Strategies (FOR US)] intervention, then answer post-intervention survey questions.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older
* Identify as Black/African- American
* Have Current or previous diagnosis of cancer
* Speak and understand English

Exclusion Criteria:

* Are younger than 18 years of age
* Do not identify as Black/African- American
* Do not have a current or previous diagnosis of cancer
* Are non - English-speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Medical Mistrust from Baseline to Post-Intervention: 12-item Group-Based Medical Mistrust Scale | Baseline and post-intervention (up to 15 minutes)
  Will assess the effect of a culturally tailored decision aid video on medical mistrust. Participants will complete the 12-item Group-Based Medical Mistrust Scale at baseline and post-intervention. This is a 12-item validated survey focused on healthcare provided in the social context of racism and discrimination. Item responses use a Likert-type scale with higher scores indicating higher agreement.
Change in Trust in Health Information from Baseline to Post-Intervention: Health Information National Trends Survey (HINTS) | Baseline and post-intervention (up to 15 minutes)
  Will assess the effect of a culturally tailored decision aid video on trust in information. Participants will complete 6 items from the National Cancer Institute - Health Information National Trends Survey (HINTS). HINTS collects nationally representative data routinely about the American public's use of cancer-related information. HINTS comprises multiple choice questions about medical research and medical records and patient-provider communications.
Change in Patient Knowledge from Baseline to Post-Intervention: Five unique question items | Baseline and post-intervention (up to 15 minutes)
  Will assess the effect of a culturally tailored decision aid video on patient knowledge about clinical trials via a five unique question items survey.
Change in Clinical Trial Participation Decision-Making Self-Efficacy from Baseline to Post-Intervention: 11-item Decision Self-Efficacy Scale | Baseline and post-intervention (up to 15 minutes)
  Will assess the effect of a culturally tailored decision aid video on clinical trial participation decision-making self-efficacy using the 11-item Decision Self-Efficacy Scale. The 11-item Decision Self-Efficacy Scale measures self-confidence or belief in one's abilities in decision making. Possible scores range from 0 to 100, with higher scores indicating more decision self-efficacy and a better outcome.
Acceptability of the intervention | At post-intervention (up to 15 minutes)
  Participants will complete a post-intervention survey to assess acceptability of the video intervention. This survey is a 5-item measure; items responded to on a Likert-type scale with higher scores indicating higher acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Vida Henderson, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/15/NCT06218615/ICF_000.pdf